CLINICAL TRIAL: NCT00254228
Title: A Clinical Study to Evaluate the Safety and Efficacy of the BrainPort™ Balance Device When Used to Improve Postural Control in Subjects With Bilateral Vestibular Disorders
Brief Title: Safety and Efficacy of the BrainPort™ Balance Device to Improve Balance in Bilateral Vestibular Hypofunction
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated due to slow recruitment
Sponsor: Wicab (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WCB1-001
Record Dates: First submitted 2005-11-10; First posted 2005-11-15 (Estimated); Last update posted 2008-10-09 (Estimated); Status verified 2008-10

CONDITIONS: Vestibular Disease
Keywords: Balance; Vestibular; Electrotactile; BrainPort; Sensory substitution; Tongue
MeSH Terms: conditions — Vestibular Diseases

INTERVENTIONS:
Device: Electrotactile sensory substitution

SUMMARY:
The purpose of this study is to determine whether the BrainPort™ balance device is safe and effective in the treatment of balance disorders in patients with Bilateral Vestibular Dysfunction.

DETAILED DESCRIPTION:
People with Bilateral Vestibular Dysfunction (BVD) often experience disabling symptoms, greatly affecting their quality of life and ability to work. Current vestibular treatment does not always allow these patients to fully recover. Many patients either do not improve or reach a plateau with conventional vestibular rehabilitation, and still have difficulty with daily function. The BrainPort™ balance device is intended to provide information about head position to the brain through electrotactile stimulation of the tongue to improve balance in subjects with vestibular disorders.

This study is a prospective, multi-center, randomized double-blinded study comparing the postural stability of BVD subjects using the BrainPort™ balance device to postural stability of control subjects using a sham device and respective baseline measures for each group. The primary objective of this study is to determine whether electrotactile stimulation of the tongue, using the BrainPort™ balance device, can improve postural stability, as measured by improvement in performance of the composite Computerized Dynamic Posturography using the NeuroCom® Sensory Organization Test in subjects with chronic bilateral vestibular dysfunction (BVD). The secondary objectives are to evaluate improvement in quality of life, as measured by the Activities Specific Balance Confidence (ABC) Scale, Dizziness Handicap Inventory (DHI), and the Dynamic Gait Index (DGI), and to demonstrate a decreased number of falls on the NeuroCom® Sensory Organization Test. In addition, we will monitor the number of falls that occur during subjects' normal activities of daily living. The long-term objective is to evaluate the safety and efficacy when the device is used over a one-year period.

ELIGIBILITY:
Inclusion Criteria:

* Documented history of acquired bilateral vestibular dysfunction for a duration of at least one year which has been unsuccessfully treated or reached a plateau with conventional vestibular rehabilitation.
* No greater than 2 successful attempts out of 6 on the NeuroCom Equitest Sensory Organization Tests 5 and 6.
* Failure on the Rotary Chair Vestibulo-ocular Reflex (VOR) Test as evidenced by a gain of less than or equal to -2 standard deviations at frequencies of .025, and .05 Hz.
* Normal corrected vision (20/40 or better).
* Able to read and understand the informed consent form, and willing to sign the informed consent form.
* Willing to complete all follow-up evaluations required by the study protocol.
* Able to stand for a period of 20 minutes in a stationary position with weight evenly distributed without moderate pain, muscle cramping or numbness in the lower extremities.

Exclusion Criteria:

* Neurological disorders other than bilateral vestibular disorder, as determined by medical history and neurological screening procedure.
* Current oral health problems as determined by health questionnaire and an examination of the oral cavity.
* Cigarette smokers and those who use chewing tobacco.
* Currently taking either benzodiazepine or barbiturate medication.
* Any medical condition as determined by the health questionnaire that would interfere with performance on the postural stability evaluation tests.
* Known neuropathies of tongue or skin tactile system.
* Peripheral neuropathies of the lower extremities.
* Prior exposure to BrainPort™ balance device (does not apply to control group subjects who cross over).
* Subjects who are unwilling or unable to adhere to all study requirements, including completion of the training period, evaluation tests, and return to clinic for a follow-up visit.
* Subjects who have undergone middle ear or other surgery with sacrifice or damage to the chorda tympani, lingual, or hypoglossal nerve.
* Subjects who have an implanted device such as a pacemaker or defibrillator.
* If the subject is female, she is pregnant.
* If the subject is unwilling to discontinue medications for dizziness or imbalance 48 hours prior to beginning the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2005-11; Study Completion 2007-12

PRIMARY OUTCOMES:
Computerized Dynamic Posturography using the NeuroCom Sensory Organization Test (SOT) composite score, taken at baseline, 1 week, 8 weeks and 12 months.

SECONDARY OUTCOMES:
Activities-specific Balance Confidence Scale (ABC)
Dizziness Handicap Inventory (DHI)
Dynamic Gait Index (DGI)
Number of falls on the NeuroCom SOT
Functional Objective Tests i.e. standing with eyes closed, on one leg, etc.
All tests taken at baseline, 1 week, 8 weeks and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Yuri P Danilov, PhD, Study Director — Wicab
Locations (5):
- United States (4):
  - Mayo Clinic, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - University of Wisconsin, Madison, Madison, Wisconsin
- Medway Balance Centre, Kent, United Kingdom

REFERENCES:
- [Background] Bach-y-Rita P, W Kercel S. Sensory substitution and the human-machine interface. Trends Cogn Sci. 2003 Dec;7(12):541-6. doi: 10.1016/j.tics.2003.10.013. PMID 14643370
- [Background] Tyler M, Danilov Y, Bach-Y-Rita P. Closing an open-loop control system: vestibular substitution through the tongue. J Integr Neurosci. 2003 Dec;2(2):159-64. doi: 10.1142/s0219635203000263. PMID 15011268
- [Background] Bach-y-rita P, Danilov YP, Tyler ME, Grimm RF. Late Human Brain Plasticity: Vestibular Substitution with a Tongue BrainPort Human-Machine Interface. Journal Intellectica, 2005 (in press).
- [Background] Bach-Y-Rita P. Emerging concepts of brain function. J Integr Neurosci. 2005 Jun;4(2):183-205. doi: 10.1142/s0219635205000768. PMID 15988797
- See also: Related Info — http://www.wicab.com